CLINICAL TRIAL: NCT01300312
Title: Evaluation of Efficacy and Tolerability of a Fixed Dose Combination of Eperisone Hydrochloride and Diclofenac Sodium in the Treatment of Acute Musculoskeletal Spasm Associated With Low Back Pain: An Observer Blind, Prospective, Randomized, Controlled Study
Brief Title: A Clinical Trial to Study the Effects of a Fixed Dose Combination of Diclofenac and Eperisone Hydrochloride With Plain Eperisone Hydrochloride in Patients With Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EIL/EPD/CT/01/2010
Record Dates: First submitted 2011-02-14; First posted 2011-02-21 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Acute Musculoskeletal Spasm Due to Low Back Pain
Keywords: eperisone; diclofenac; low back pain
MeSH Terms: conditions — Low Back Pain | interventions — eperisone; Diclofenac

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Eperisone hydrochloride and Diclofenac sodium
- 2 (Active Comparator)
  Interventions: Drug: Eperisone hydrochloride

INTERVENTIONS:
Drug: Eperisone hydrochloride and Diclofenac sodium — Fixed dose capsule formulation of eperisone hydrochloride 50 mg plus diclofenac sodium 50 mg to be given 3 times a day after meals for 7 to 10 days
  Arms: 1
Drug: Eperisone hydrochloride — eperisone hydrochloride 50 mg as tablet formulation to be given 3 times daily after meals for 7 to 10 days
  Arms: 2

SUMMARY:
The purpose of this study is to investigate the effects of a fixed dose combination of diclofenac and eperisone hydrochloride compared with plain eperisone hydrochloride in patients with low back pain.

DETAILED DESCRIPTION:
This study is an observer-blind, prospective randomized, controlled study to evaluate efficacy and safety of fixed dose combination of eperisone hydrochloride 50 mg and diclofenac sodium 50 mg three times daily with plain eperisone hydrochloride 50 mg three times daily in patients with musculoskeletal spasm associated with low back pain. A total of 240 adult patients of either sex, 120 patients in each arm, who fulfill the inclusion and exclusion criteria will be included in this study. The patients will be evaluated at Days 3, 7 and 10 of the study visit for efficacy and safety. The efficacy evaluation includes objective parameters like Finger-to-Floor distance, Lasegue's sign, tenderness of par vertebral muscles, lumbar and dorsal hypermyotonia, leg tendon reflexes, need for rescue medication and subjective parameters like improvement in lumbar cinesalgia, pain in lower extremities, sensory disturbances of lower limb, and Global Assessment of Response to Therapy (PGART). Patients will be evaluated for safety on the clinical adverse events reported during the study period, sedation on drowsy alert scale and Global Assessment of Tolerability to Therapy (PGATT). The patients will also be evaluated for laboratory safety as assessed by measuring laboratory parameters for hemogram, renal and hepatic parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patient of either sex between 18 to 60 years of age
* Patients with confirmed diagnosis of Acute Musculoskeletal spasm with Low

Back Pain due to any of the following causes:

1. Spondylosis deformans
2. Prolapsed Intervertebral Disc (PID)
3. Muscle Sprains with spasms

   * Patients willing to take the medications as directed and willing to come for the follow-ups
   * Willing to comply with the protocol requirements
   * Willing to give the written informed consent

Exclusion Criteria:

* Patients associated with other lumbar spinal tract conditions such as spondylitis, fracture, cancers, severe arthritis and osteoporosis.
* Muscular diseases such as myositis, poliomyelitis, muscular dystrophy and myotonia.
* Other known systemic diseases affecting the neurological or endocrine.
* Patients with moderate to severe hepatic impairment (defined as increase in serum bilirubin, serum glutamic oxaloacetic transaminase (SGOT) and serum glutamic pyruvic transaminase (SGPT) by >2.5 times the upper reference level of the laboratory values) and renal impairment (defined as increase in serum creatinine and Blood urea nitrogen by >2.5 times the upper reference level of the laboratory values).
* Patients who had taken any form of skeletal muscle relaxant in the previous 7 days.
* Pregnant / Lactating woman or women of child bearing potential not following adequate contraceptive measures.
* Patients with known hypersensitivity to ingredients of study/active comparators.
* Patients with any previous history of or current episode of cardio-vascular disorders.
* Subject known to be having any of the following disorder: renal failure, bulimia, hypo and hyperthyroidism, nephrotic syndrome, anorexia nervosa, biliary obstruction, severe cardiac dysfunction.
* Uncontrolled diabetes mellitus or any other metabolic disorder.
* Pediatric and pregnant patients.
* Patients with history of alcoholic/substance abuse.
* Treatment with any investigational drug in the preceding 4 weeks.
* Patients with active or recent history of, inflammatory diseases of the gastrointestinal tract such as peptic ulcer, gastritis, regional enteritis, or ulcerative colitis.
* Patients in whom acetylsalicylic acid (ASA) or other non-steroidal anti-inflammatory agents (NSAIDs) have induced asthma, rhinitis, urticaria or other allergic manifestations.
* Any other condition that, in the opinion of the investigator, does not justify the inclusion of the subject in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 239 (Actual)
Dates: Start 2011-02; Primary Completion 2011-06 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Finger to Floor Distance: Improvement in Finger to Floor Distance compared to baseline. | Day 1,3,7 and 10 of study period
  Improvement in the Fingertip-to-Floor-surface Distance [FFD] from baseline on Day 3, Day 7 & Day 10. Finger Floor Distance [FFD] is an index for the mobility of the lumbar spinal cord and is measured as the distance between the finger-tip of the middle Finger to the Floor-surface as determined while standing with the spinal cord flexed with complete extension of knee joint. It is measured in millimeters.

SECONDARY OUTCOMES:
Objective Efficacy Assessment: Improvement in Lasegue's sign compared to baseline | Day 1, 3, 7 and 10 of study period
  Lasegue's sign is the lumbar pain [or exacerbation of existing pain] experienced by the patient on passive movement of the legs during flexion of hip joint i.e. passive straight leg raising. It is assessed as either 'Positive' or 'Negative' sign.
Subjective Efficacy Assessment: Improvement of lumbar cinesalgia compared to baseline | Day 1, 3, 7 and 10 of study period
  Improvement in Lumbar Cinesalgia (pain in lumbar region) assessed on a 0 to 100mm Visual Analogue Scale (VAS) with '0' representing 'NO PAIN' and 100 representing 'SEVERE INTOLERABLE PAIN'

CONTACTS AND LOCATIONS:
Overall Officials: Suyog Mehta, Study Director — General Manager - Medical and Regulatory Affairs, Eisai Pharmaceuticals India Private Limited
Locations (4):
- India (4):
  - Department of Orthopedics, Government Medical College, Aurangabad, Maharashtra
  - Deore Hospital, Aurangabad, Maharashtra
  - Department of Orthopedics, Grant Medical College and Sir J.J. Group of Hospitals, Mumbai, Maharashtra
  - Kabre Orthopedic, Spine & Dental Care, Pune, Maharashtra